CLINICAL TRIAL: NCT07208292
Title: Real-world Study on Preoperative Application of Rezvilutamide
Acronym: RWS-GU001
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pudong New Area Gongli Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GLYY1s2025-040; mierxiati@fudan.edu.cn (Other: Shanghai Pudong New Area Gongli Hospital)
Record Dates: First submitted 2025-07-23; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Preoperative Evaluation
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Prostate Specimens Removed by Surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Real-world study on Preoperative Application of Rezvilutamide

DETAILED DESCRIPTION:
Observation on Postoperative and Long-term Indicators of Rezvilutamide in Perioperative Medication, Including Postoperative Pathological Complete Response Rate, Postoperative Biochemical Recurrence, etc.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation: Confirmed as prostate adenocarcinoma by ultrasound/MRI-guided prostate biopsy, with ISUP grade ≥ 2 (Gleason score ≥ 7);
* Clinical staging (based on AJCC 8th edition):High-risk localized: cT3a or PSA > 20 ng/ml or Gleason score ≥ 8;Locally advanced: cT3b-4 or positive pelvic lymph nodes (cN1);
* Surgical feasibility: Multidisciplinary team (MDT) assessment considers that R0/R1 resection can be achieved;
* Laboratory requirements:Hemoglobin ≥ 90 g/L, platelets ≥ 100×10^9/L;Liver function: ALT/AST ≤ 2.5×ULN, bilirubin ≤ 1.5×ULN;Renal function: eGFR ≥ 30 mL/min/1.73m².

Exclusion Criteria:

* Disease-related: Distant metastasis (M1, including bone metastasis or visceral metastasis);Pathology indicating neuroendocrine differentiation or small cell carcinoma component > 10%;
* Treatment-related:Previous history of receiving radiotherapy, cryotherapy, or systemic chemotherapy for prostate cancer;History of other malignant tumors within 5 years (except non-melanoma skin cancer);
* Comorbidities: Uncontrolled cardiovascular diseases (e.g., NYHA Class III heart failure, myocardial infarction within 6 months);History of severe epilepsy (requiring long-term use of anticonvulsant drugs);・Others:Known allergy to relugolix or LHRH analogs;Participation in other interventional clinical trials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A description of the population from data from Postoperative Patients with Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response（PCR） | Postoperative Immediate Pathological Diagnosis
  A pathological complete response (pCR) signifies the complete absence of detectable invasive cancer cells in tissue surgically removed from a patient. This evaluation is made by a pathologist after a patient has undergone neoadjuvant therapy-a course of treatment before their primary surgery.
Minimal Residual Disease(MRD) | Postoperative Immediate Pathological Diagnosis
  Minimal residual disease is that not detected by conventional imaging studies and clinically the patient remains disease free. However, with time these dormant cells will awaken and disease progression occurs, resulting in clinically and radiological detectable metastatic disease.
Biochemical Recurrence(BCR) | through study completion, an average of 2 year
  Biochemical recurrence in prostate cancer is one in which rising serum prostate-specific antigen (PSA) levels point to the existence of disease,PSA>0.2ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Mierxiati Abudurexiti, Study Chair — Shanghai Pudong New Area Gongli Hospital

IPD SHARING:
Plan to Share IPD: No